CLINICAL TRIAL: NCT01536834
Title: A Pilot Clinical Investigation in Adults to Evaluate the Safety and Performance of a Class IIa Medical Device for the Treatment of Plantar Warts (Verrucas)
Brief Title: Safety & Performance Study of Verruca Treatment Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPD396 02
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2012-02

CONDITIONS: Verruca; Plantar Wart
Keywords: Verruca; Plantar Wart; Medical Device; Podiatry; Footcare
MeSH Terms: conditions — Warts | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Device (Experimental): The Investigational device is a liquid in a delivery system for the treatment of verrucas
  Interventions: Device: Medical Device

INTERVENTIONS:
Device: Medical Device

SUMMARY:
This is a non comparative pre-CE marking pilot clinical investigation is required to evaluate the safety and performance in intended use of the Verruca treatment - NPD396, Class IIa medical device for verrucas in the adult population. The treatment regime will be topical application of the Verruca treatment to the verruca, identified as the reference, once daily for 4 weeks.

Patient & investigator derived outcomes will also be collected to assess clinical performance and adverse events and adverse device effects will be reported to assess safety profile.

Patient assessments will take place pre-treatment to determine patient demography, baseline clinical status, pain and verruca size prior to treatment. Compliance with treatment schedule will be collected via patient diary cards. Furthermore, patients will be assessed on day 2 after starting treatment and then again at 7, 14, 21 & 28 days after starting treatment. Diary cards will completed through-out the investigation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >18 years
* Patients with verrucas
* Patients should be willing to take part, able to understand the information given to them and give written consent

Exclusion Criteria:

* Patient with more than two areas affected by verrucas on one foot
* Patient who are actively treating or have treated their wart within the past 8 weeks
* Patient suspected to be immunocompromised or are taking immunosuppressants
* Patient who suffer from impaired feeling due to diabetes, peripheral vascular disease or neuropathy.
* Current participation in another clinical investigation or participation within the last 30 days.
* Patient with known sensitivity/allergies to the test materials or any of their ingredients.
* Significant current or past medical history of hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, locomotor or psychiatric disease, which, in the opinion of the Investigator, would compromise the safety of the volunteer or affect the outcome of the investigation (as determined from self-reported medical history questionnaire).
* Patient in a situation which in the view of the investigator could interfere with optimal participation in the investigation or constitute a special risk for these patients.
* Patient who scar easily or are prone to hypertrophic or Keloid scarring.
* Patient who have previously had an unfavourable reaction to any products for the feet and which involved swelling of the foot, or a requirement for painkillers or antibiotics.
* Pregnant and lactating females, or those actively seeking to become pregnant in the next month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint | 4 weeks
  Safety will be assessed in terms of severity, frequency and seriousness of any complications, adverse events or adverse device effects.

SECONDARY OUTCOMES:
Efficacy endpoint presence/absence of verruca by podiatrist | 4 weeks
  Presence (& Area) or absence of verruca at each visit, as determined by podiatrist using photographic data.
Efficacy endpoint presence/absence of verruca and pain by patient | 4 weeks
  Patient's assessment of presence or absence of the verruca and associated pain during follow-up period using VAS within diary cards. A set of Patient perception questions will also be included in the diary card.

CONTACTS AND LOCATIONS:
Locations (1):
- Mr. Andrew Ryals, Wakefield, Yorkshire, United Kingdom